CLINICAL TRIAL: NCT00082966
Title: A Phase II Study of PS-341 (Bortezomib) in Patients With Relapsed or Refractory Hodgkin's Lymphoma
Brief Title: Bortezomib in Treating Patients With Relapsed or Refractory Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01812; CALGB-50206; CDR0000361745; U10CA031946 (NIH)
Record Dates: First submitted 2004-05-14; First posted 2004-05-17 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2013-06

CONDITIONS: Adult Lymphocyte Depletion Hodgkin Lymphoma; Adult Mixed Cellularity Hodgkin Lymphoma; Adult Nodular Sclerosis Hodgkin Lymphoma; Recurrent Adult Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — tanespimycin; Bortezomib

ARMS (1):
- Arm I (Experimental): Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 8 courses in the absence of rapid disease progression or unacceptable toxicity.
  Interventions: Drug: 17-N-allylamino-17-demethoxygeldanamycin/bortezomib

INTERVENTIONS:
Drug: 17-N-allylamino-17-demethoxygeldanamycin/bortezomib — Given IV

SUMMARY:
Phase II trial to study the effectiveness of bortezomib in treating patients who have relapsed or refractory Hodgkin's lymphoma. Bortezomib may stop the growth of cancer cells by blocking the enzymes necessary for their growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of bortezomib in patients with relapsed or refractory Hodgkin's lymphoma using overall response rate as the primary efficacy endpoint.

II. To assess time to progression and 2-year overall survival after bortezomib therapy.

III. To evaluate the safety and tolerability of bortezomib in patients with relapsed/refractory Hodgkin's lymphoma.

OUTLINE: This is a multicenter study.

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 8 courses in the absence of rapid disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed classical Hodgkin's lymphoma

  * No bone marrow biopsies or fine needle aspirates as the sole means of diagnosis
  * Core biopsies allowed if they contain adequate tissue for primary diagnosis
* The following subtypes are allowed:

  * Nodular sclerosis
  * Lymphocyte rich
  * Mixed cellularity
  * Lymphocyte depletion
  * Classical Hodgkin's lymphoma, not otherwise specified
* No nodular lymphocyte-predominant Hodgkin's lymphoma
* Relapsed or refractory disease after at least 1 prior standard systemic cytotoxic chemotherapy regimen
* Measurable disease by physical exam or imaging studies

  * Any tumor mass > 1 cm is allowed
  * No non-measurable disease only, including the following:

    * Bone lesions
    * Ascites
    * Pleural or pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Bone marrow
* No curative option available with high-dose therapy and stem cell transplantation
* Performance status - 0-2
* Absolute neutrophil count ≥ 750/mm^3
* Platelet count ≥ 75,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST ≤ 2.5 times ULN
* Creatinine ≤ 2.5 mg/dL
* No sensory or motor peripheral neuropathy ≥ grade 2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for up to 3 months after study participation
* See Disease Characteristics
* Prior stem cell transplantation allowed
* See Disease Characteristics
* No concurrent chemotherapy
* No concurrent dexamethasone or other steroidal antiemetics

  * Concurrent steroids for adrenal failure allowed
* Concurrent hormonal therapy for non-disease related conditions (e.g., insulin for diabetes) allowed
* Prior radiotherapy to a symptomatic lesion or one that may produce disability (e.g., unstable femur) is allowed provided other measurable disease is present
* No concurrent palliative radiotherapy
* Recovered from all prior treatment
* No prior bortezomib or other proteosome inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-03; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Up to 3 years
Time to progression | Up to 5 years
Overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Bartlett, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States